CLINICAL TRIAL: NCT05092425
Title: Analysis of Risk Factors for Children With Heterochronous Indirect Hernia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Hospital (Other)
Collaborators: Children's Hospital of Hebei Province (Other); Shengjing Hospital (Other); Children's Hospital of Nanjing Medical University (Other); Anhui Provincial Children's Hospital (Other); Tianjin Children's Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Tongji Hospital (Other); Zunyi Medical College (Other); Maternal and Child Health Hospital of Henan Province (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021R076
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Inguinal Hernia, Direct; Child, Only; Laparoscopic Surgery
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with CPPV: Group 1 is childrens with contralateral patent processus vaginalis.
- without CPPV: Group 2 is childrens without contralateral patent processus vaginalis.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention
  Groups: without CPPV

SUMMARY:
Laparoscopic contralateral patent processus vaginalis (CPPV) repair in infancy and childhood is still debatable, due to the high CPPV rate but low contralateral metachronous hernia (MCIH) rate. In order to found risk factors for MH, we conducted this prospective study.

This is an multi-center investigator-initiated observational prospective trial. After informed all the benefits and risks of repair CPPV simultaneously, those patients with unilateral inguinal hernia whose parents preferred not to repair CPPV simultaneously will be assigned in the study. All information about demographic data, hernia side, CPPV type and CPPV diameter will be recorded. The subjects will be followed up until MCIH developing or to 24 months postoperatively. Patients will be analyzed to identify the risk factors for MH.

DETAILED DESCRIPTION:
Inguinal hernia (IH) is one of the most common diseases in pediatric surgery with an overall rate of 0.8-4.4%1, and 75-90% of these patients were with unilateral inguinal hernia (UIH). Children with UIH have a chance of subsequently developing metachronous contralateral inguinal hernia (MCIH). Whether to explore the contralateral side in children with UIH has been debated for many decades. Surgeons used to practiced contralateral exploration in children due to the high reported incidence of a contralateral patent processus vaginalis (CPPV) and the increased risk of general anesthesia at the very young. Then surgeons noted that only few CPPV might develop into a clinical hernia, and routine exploration puts both testicles and both vas deferens at risk. Because of this fact, many surgeons have abandoned routine contralateral exploration.

As laparoscopic hernia repair is performed in children, CPPV exploration and ligation become much easier, without extra incision. A lot of literature reported that CPPV ligation could prevent MCIH and regarded this as a major benefit of laparoscopic hernia repair. Still, the laparoscopic CPPV rates (28%-66%) are much higher than the rates of MCIH developing (2.4% to 13.9%). Therefore one would need to perform 4 to 21 operations to prevent one future hernia. Whether to close the CPPV simultaneously in children with UIH is still controversial. We think that either yes or no is not the best answer. It is essential to identify the risk factors of MCIH to make the best strategies to balance the risks and benefits. We, therefore, designed a prospective observational study of pediatric patients with UIH to detect the risk factors of MCIH.

This is an multi-center investigator-initiated observational prospective trial. After informed all the benefits and risks of repair CPPV simultaneously, those patients with unilateral inguinal hernia whose parents preferred not to repair CPPV simultaneously will be assigned in the study. Patients included in this trial will receive laparoscopically extraperitoneal high ligation of the hernia sac and detection of the contralateral side. All information about demographic data, hernia side, CPPV type and CPPV diameter will be recorded. The subjects will be followed up until MCIH developing or to 24 months postoperatively. Patients will be analyzed to identify the risk factors for MH.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral indirect inguinal hernia in males and females (0-18 years old)
* Healthy (based on history), non-athletes
* The guardian understands the purpose and risks of the study and signs the relevant informed consent

Exclusion Criteria:

* Recurrent indirect inguinal hernia
* Incarcerated indirect inguinal hernia
* The ultrasonography shows contralateral patent processus vaginalis
* with other systemic diseases (such as chronic constipation, chronic cough, cardiopulmonary insufficiency, liver and kidney insufficiency, abdominal wall malformation, urinary tract malformation, etc.)

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Childrens dianosed as unilateral indirect inguinal hernia in Out-patient with a healthy history, non athelets. And parents preferred not to repair CPPV simultaneously in Laparoscopic indirect inguinal hernia repairing after informed all the benefits and risks
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The rate of MCIH | 08.01.2021-07.31.2021
  the rate of MCIH developments after 24 months

SECONDARY OUTCOMES:
Complications | 08.01.2021-07.31.2024
  hernia recurrances, and postoperative complications such as wound infection, scrotal edema, haematoma, testicular atrophy, and iatrogenic cryptorchidism.

CONTACTS AND LOCATIONS:
Overall Officials: Zhibao Lv, PhD, Study Chair — Shanghai Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kokorowski PJ, Wang HH, Routh JC, Hubert KC, Nelson CP. Evaluation of the contralateral inguinal ring in clinically unilateral inguinal hernia: a systematic review and meta-analysis. Hernia. 2014 Jun;18(3):311-24. doi: 10.1007/s10029-013-1146-z. Epub 2013 Aug 21. PMID 23963735
- [Background] Dreuning K, Maat S, Twisk J, van Heurn E, Derikx J. Laparoscopic versus open pediatric inguinal hernia repair: state-of-the-art comparison and future perspectives from a meta-analysis. Surg Endosc. 2019 Oct;33(10):3177-3191. doi: 10.1007/s00464-019-06960-2. Epub 2019 Jul 17. PMID 31317333
- [Background] Nakashima M, Ide K, Kawakami K. Laparoscopic versus open repair for inguinal hernia in children: a retrospective cohort study. Surg Today. 2019 Dec;49(12):1044-1050. doi: 10.1007/s00595-019-01847-0. Epub 2019 Jul 16. PMID 31312986
- [Background] Kantor N, Travis N, Wayne C, Nasr A. Laparoscopic versus open inguinal hernia repair in children: which is the true gold-standard? A systematic review and meta-analysis. Pediatr Surg Int. 2019 Sep;35(9):1013-1026. doi: 10.1007/s00383-019-04521-1. Epub 2019 Jul 10. PMID 31292721
- [Background] Shaughnessy MP, Maassel NL, Yung N, Solomon DG, Cowles RA. Laparoscopy is increasingly used for pediatric inguinal hernia repair. J Pediatr Surg. 2021 Nov;56(11):2016-2021. doi: 10.1016/j.jpedsurg.2021.01.032. Epub 2021 Jan 27. PMID 33549307
- [Background] Li Y, Wu Y, Wang C, Wang Q, Zhao Y, Ji Y, Xiang B. Incidence of pediatric metachronous contralateral inguinal hernia and the relationship with contralateral patent processus vaginalis. Surg Endosc. 2019 Apr;33(4):1087-1090. doi: 10.1007/s00464-018-6359-x. Epub 2018 Sep 25. PMID 30255331
- [Background] Matsuda A, Miyashita M, Matsumoto S, Sakurazawa N, Kawano Y, Kuriyama S, Sekiguchi K, Ando F, Matsutani T, Uchida E. Laparoscopic transabdominal preperitoneal repair for strangulated inguinal hernia. Asian J Endosc Surg. 2018 May;11(2):155-159. doi: 10.1111/ases.12438. Epub 2017 Oct 19. PMID 29052338
- [Background] Zhu LL, Xu WJ, Liu JB, Huang X, Lv ZB. Comparison of laparoscopic hernia repair and open herniotomy in children: a retrospective cohort study. Hernia. 2017 Jun;21(3):417-423. doi: 10.1007/s10029-017-1607-x. Epub 2017 Apr 19. PMID 28424930
- [Background] Zhao J, Chen Y, Lin J, Jin Y, Yang H, Wang F, Zhong H, Zhu J. Potential value of routine contralateral patent processus vaginalis repair in children with unilateral inguinal hernia. Br J Surg. 2017 Jan;104(1):148-151. doi: 10.1002/bjs.10302. Epub 2016 Oct 25. PMID 27778329
- [Background] Ahmed H, Youssef MK, Salem EA, Fawzi AM, Desoky EA, Eliwa AM, Sakr AM, Shahin AM. Efficacy of laparoscopically assisted high ligation of patent processus vaginalis in children. J Pediatr Urol. 2016 Feb;12(1):50.e1-5. doi: 10.1016/j.jpurol.2015.05.036. Epub 2015 Sep 15. PMID 26421498
- [Background] Esposito C, Escolino M, Turra F, Roberti A, Cerulo M, Farina A, Caiazzo S, Cortese G, Servillo G, Settimi A. Current concepts in the management of inguinal hernia and hydrocele in pediatric patients in laparoscopic era. Semin Pediatr Surg. 2016 Aug;25(4):232-40. doi: 10.1053/j.sempedsurg.2016.05.006. Epub 2016 May 11. PMID 27521714